CLINICAL TRIAL: NCT06634316
Title: Nutritional Management of Sarcopenia in Patients With Heart Failure
Brief Title: Sarcopenia in Patients With Heart Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Insuficiencia cardiaca 2
Record Dates: First submitted 2023-08-23; First posted 2024-10-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Diet, Mediterranean; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mediterranean diet (Active Comparator): Mediterranean diet and physical exercise
  Interventions: Other: Mediterranean diet; Combination Product: Vitamin D supplementation; Combination Product: Physical exercise
- Standard hypercaloric hyperproteic Oral supplement (Experimental): Standard hypercaloric hyperproteic oral supplement plus Mediterranean diet and physical exercise
  Interventions: Other: Mediterranean diet; Dietary Supplement: Hypercaloric, hyperproteic oral nutritional supplement; Combination Product: Vitamin D supplementation; Combination Product: Physical exercise
- Protein module (Experimental): Protein module (10g/day) plus Mediterranean diet and physical exercise
  Interventions: Other: Mediterranean diet; Dietary Supplement: Protein module; Combination Product: Vitamin D supplementation; Combination Product: Physical exercise

INTERVENTIONS:
Other: Mediterranean diet — Mediterranean diet recommendations and daily physical exercise
Dietary Supplement: Hypercaloric, hyperproteic oral nutritional supplement — Hypercaloric, hyperproteic oral supplement combined with Mediterranean diet recommendations (2 per day) and daily physical exercise
  Arms: Standard hypercaloric hyperproteic Oral supplement
Dietary Supplement: Protein module — Protein module (10g/day) combined with Mediterranean diet recommendations and daily physical exercise
  Arms: Protein module
Combination Product: Vitamin D supplementation — Calcifediol supplement administered orally in order to reach sufficiency levels (30 ng/ml)
Combination Product: Physical exercise — Physical exercise adapted to patients with heart failure (Cardiac rehabilitation)

SUMMARY:
Sarcopenia is a frequent complication in patients with cancer and chronic diseases, it is characterized by decreased muscle strength and fatigue due to reduced skeletal muscle mass, which is accompanied by atrophy and decreased quality of muscle tissue. In all cases, it negatively impacts treatment tolerance, clinical outcomes and survival, in consequence, quality of life of these patients decreases while morbidity, mortality and costs increase. In this context, appropriate nutritional screening and early nutrition support are extremely recommended, to this aim, in some cases, oral nutritional supplements (ONS) are necessary; ONS could have a standard formula or be enriched with specific nutrients. There is a lack of evidence for supporting its use or the use of protein modules in other clinical conditions including patients with heart failure

ELIGIBILITY:
Inclusion Criteria:

* Patients with a previous admission due to HF in the previous 12 months
* Moderate or severe LVEF
* Both sexs
* Age >18 years old.

Exclusion Criteria:

* MDRD <15 ml/min
* End-stage liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | 6 months
  Changes in muscle mass
Functionality | 6 months
  Changes in functionality determined by the up and go test

SECONDARY OUTCOMES:
Albumin | 6 months
  Changes in serum albumin levels (g/dl)
C-RP | 6 months
  Changes in serum C-RP (g/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- IMIBIC, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided